CLINICAL TRIAL: NCT01009437
Title: A Phase I/II Trial of Short Course Pre-Operative Ritonavir To Determine Akt Inhibition in Breast Cancer
Brief Title: Ritonavir and Its Effects on Biomarkers in Women Undergoing Surgery for Newly Diagnosed Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008NTLS083; UMN-0809M45461 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Breast Cancer
Keywords: HER2-negative breast cancer; HER2-positive breast cancer; estrogen receptor-positive breast cancer; triple-negative breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; ductal breast carcinoma in situ
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating | interventions — Ritonavir; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control Arm - No Ritonavir (Active Comparator): Five ER+, HER2- breast cancer patients meeting all study eligibility will be enrolled prior to the start of phase I recruitment to act as controls (no ritonavir will be given-will receive therapeutic conventional surgery) to confirm that anesthesia does not affect EET levels. Core biopsies, surgical tumor/normal tissue and pre- and post- surgery blood samples will be collected for comparison with the treatment group.
  Interventions: Procedure: therapeutic conventional surgery
- Ritonavir - Escalating Doses (I) (Experimental): Standard phase I dose escalation (with therapeutic conventional surgery) will be used with 3 levels of ritonavir given - 200 mg bid, 400 mg bid, and 600 mg bid for the following groups:
  1. ER+, HER2-
  2. ER+, HER2+
  3. ER-, HER2+
  4. ER-, PR+, HER2-
  5. ER-, PR-, HER2-
  Interventions: Drug: ritonavir; Procedure: therapeutic conventional surgery
- Ritonavir - Maximum Tolerated Dose (II) (Experimental): Phase II: Once the maximum tolerated dose (MTD) of ritonavir is established, 19 ER+, HER2- patients will be enrolled at MTD during the phase II component along with therapeutic conventional surgery.
  Interventions: Drug: ritonavir; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Drug: ritonavir — Phase I: Dose escalation will be used with 3 levels of ritonavir given - 200 mg twice a day (bid), 400 mg bid, and 600 mg bid.
  Phase II: Dose will be maximum tolerated dose from Phase I.
  Other Names: NORVIR® tablets
  Arms: Ritonavir - Escalating Doses (I); Ritonavir - Maximum Tolerated Dose (II)
Procedure: therapeutic conventional surgery — Tissue collection is from all patients, including the control, phase I and phase II patients.
  Other Names: Surgery

SUMMARY:
RATIONALE: Ritonavir may stop the growth of tumor cells by blocking some of the enzymes needed for cancer cell growth. Studying samples of blood and tissue from patients with breast cancer in the laboratory may help doctors learn more about the effects of ritonavir on biomarkers involved in breast cancer growth.

PURPOSE: This phase I/II trial is studying the best dose of ritonavir and its effects on biomarkers in women undergoing surgery for newly diagnosed breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effects of ritonavir on Akt activity, UPR, Ki67 LI, and ROS in a triple-negative breast cancer model.
* Determine the maximum tolerated dose of ritonavir in women with newly diagnosed breast cancer. (Phase I - enrollment complete)

OUTLINE: This is a multicenter, phase I dose-escalation study followed by a phase II study. *Note: This trial never moved forward to Phase ll.

Control Group - Five patients with estrogen receptor positive (ER+) and human epidermal growth factor 2 negative (HER2-) breast cancer are enrolled before the start of phase I recruitment.

Phase I Group - Twelve breast cancer patients with either 1)ER+, HER2-, or 2)ER+, HER2+, or 3) ER-, HER2+, or 4) ER-, PR+, HER2-, or 5) ER-, PR-, HER2- will be enrolled for dose escalation study.

Phase II Group - Nineteen ER+, HER2- patients will be enrolled for ritonavir pharmacokinetic study after maximum tolerated dose (MTD) is established.

* Control: Patients do not receive ritonavir.
* Phases I and II: Patients receive oral ritonavir twice daily for 5 days in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery as deemed appropriate by the surgeon and based on patient preference (mastectomy or lumpectomy with sentinel node procedure and/or axillary node dissection).

All patients undergo blood and tissue sample collection periodically for biomarker research studies. Samples from patients enrolled in the control group are compared with the samples from patients enrolled in phase I and II.

ELIGIBILITY:
Inclusion criteria:

* Newly diagnosed biopsy proven breast cancer for which a lumpectomy or mastectomy is planned.

  * Control Selection
* ER+, HER2-: estrogen receptor positive (ER+) and human epidermal growth factor receptor 2 negative (HER2 -) as defined according to institutional standards.

  * Phase I Selection
* ER+, HER2-
* ER+, HER2+
* ER-, HER2+
* ER-, PR+, HER2-
* ER-, PR-, HER2-

  * Phase II Selection
* ER+HER2-: as defined for controls Menstrual status will be noted as either pre- or postmenopausal. For the purpose of this study, postmenopausal is defined as no menstrual period for 12 months or longer or bilateral oophorectomy
* Sufficient tumor tissue from the diagnostic core biopsy, either as a block or a minimum of 5 slides
* Tumor must be greater than 1 centimeter as measured by clinical exam, mammogram, ultrasound or MRI. - No prior treatment for breast cancer in the affected breast.
* Karnofsky performance status >70%
* No prior treatment for breast cancer in the affected breast
* Adequate organ function for receiving study drug within 14 days 1st dose of study drug
* Women of childbearing potential are required to use an effective method of contraception
* Voluntary written consent

Exclusion criteria:

* Pregnant or lactating.
* Known positive HIV status or on medications for HIV
* Diagnosis of diabetes due to potential problems with insulin resistance and hyperglycemia
* Any pre-existing gastrointestinal complaints including nausea, abdominal pain and/or diarrhea
* Known hypersensitivity to ritonavir or any of the tablet ingredients
* Co-administration of ritonavir is contraindicated with any of the drugs - Contraindicated Drugs because competition for primarily CYP3A by ritonavir could result in inhibition of the metabolism of these drugs and create the potential for serious and/or life-threatening reactions such as cardiac arrhythmias, prolonged or increased sedation, and respiratory depression. Voriconazole is an exception in that co-administration of ritonavir and voriconazole results in a significant decrease in plasma concentrations of voriconazole. If the patient cannot discontinue a contraindicated drug, she is not eligible for the trial.
* Incompatible Drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-05-26 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Inhibition of breast cancer by targeting Hsp90-Akt pathway | Pre and Post Treatment

SECONDARY OUTCOMES:
Activation of apoptosis markers | Pre and Post Treatment
Modulation of autophagy markers | Pre and Post Treatment
Alteration of plasma levels of eicosanoids | Pre Treatment and 3 Hours Post Treatment
Induction of Hsp70 in peripheral blood mononuclear cells | Pre Treatment and 3 Hours Post Treatment
Reduction of ERα in ERα+ tumors | Pre and Post Treatment
Changes in TNF-α and IL-6 levels as well as reduction in intratumoral nuclear NF-kB and phospho-Stat3 | Pre and Post Treatment
Alteration of urine eicosanoid levels | Pre and Post Treatment
Alteration of plasma and urine eicosanoid levels resulting from tumor resection. | Pre and Post Treatment
Induction of the unfolded protein response (UPR) assayed by grp78 or related markers (phospho-PERK, ATF-4, and CHOP) | pre- and post-surgery
inhibition of tumor growth markers (Ki67 LI, Hsp90, phosphorylated AKT) | pre- and post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: David A. Potter, M.D., Ph.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (2):
- United States (2):
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota
  - The Kimmel Cancer Center at Jefferson University, Philadelphia, Pennsylvania